CLINICAL TRIAL: NCT03958539
Title: Prevention of Primary Foot Ulcers in High-risk Diabetes Patients (PrOFoUnD): a Cluster Randomised Trial of 3D Printed Insoles Versus Standard Care
Brief Title: Prevention of Primary Foot Ulcers in High-risk Diabetes Patients
Acronym: PROFOUND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding during the pandemic
Sponsor: Countess of Chester NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other); Staffordshire University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 265590; 265590 (Other: IRAS)
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus; Foot Ulcer, Diabetic; Primary Prevention
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: As this study involves a complex intervention in the form of a pathway, we chose a cluster randomisation design to mitigate the risk of contamination across the groups. The podiatry units will find it much easier to follow one pathway for all participants in their sites. We also reduce the cost by halving the number of foot scanners required to be purchased (and the staff training required) for the study by using cluster randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): 6 sites out of a total of 12 will act as the intervention sites. 450 Patients with high risk of primary DFUs defined by peripheral sensory neuropathy and callus formation or critical limb ischaemia or on renal replacement therapy will be cluster randomised to be provided with bespoke 3-D printed insoles.
  Interventions: Device: 3D printed insoles for normal footware
- Control (No Intervention): 6 sites out of a total of 12 will act as the control sites providing standard care. 450 Patients with high risk of primary DFUs defined by peripheral sensory neuropathy and callus formation or critical limb ischaemia or on renal replacement therapy will be cluster randomised to standard care

INTERVENTIONS:
Device: 3D printed insoles for normal footware — Imprints are low-cost, bespoke, 3D-printed orthotics designed to prevent diabetic foot ulceration by redistributing and lowering peak foot pressures. This is achieved by using different density zones designed specifically for the patient. The patient's foot shape and pressure zone are capture by a 3D imaging system. Once scanned the software automatically identifies the peak pressure zones, matches these with the correct material and stiffness (densities), fits the insole arch to the patient and generates the insole.
  The imprints insole is divided into four pressure zones: heel, midfoot, metatarsal head region and toes. These zones are printed with different stiffness to account for the difference in loading between them. The design of the pressure zones is automatically matched to the shape of each individual foot with the help of the 3D scan.
  Arms: Intervention arm

SUMMARY:
This is a primary prevention study which aims to assess reduction in the rate of diabetic foot ulcers in patients with high-risk diabetic feet using 3D printed insoles compared to standard care

DETAILED DESCRIPTION:
Once a patient with diabetes develops a foot ulcer 80% are likely to have a lower limb amputation in the future. Amputation carries a considerable burden of cost and impaired quality of life (QOL) and is associated with a 5-year mortality rate of 70%. Once a patient develops an ulcer they remain at high risk for life and are likely to suffer considerable morbidity, debilitation, reduced quality of life and numerous attendances with health care professionals including emergency hospital presentation. There are significant costs associated with the management of diabetes foot ulcers (DFU) which accounts for £1 billion of NHS funding and an average weekly care cost of £208 per person. Both diabetes ulcers and amputation for the most part are preventable providing that patients have effective glycaemic control, regular foot assessments, care for their feet appropriately and wear appropriate footwear or orthotic wear to prevent ulceration.

The focus of this initiative is to utilise digital capability by 3D scanning systems in the community for the provision of highly cost-effective 3D printed soles for shoes which distribute the pressure on the feet whilst having the flexibility of being used in general footwear, thus improving compliance. The cost of these soles is very low at approximately £40 for two pairs. More complex orthotics cost on average £525 each. Scanners and software are likely to be offered free if this is scaled up. The investigators are proposing to work closely with podiatrists in local foot protection services to assess a number of patients at high risk of foot ulcer and deliver a care bundle, which will include assessment, education around both foot care and promoting structured education and 3D sole provision.

The study aims to assess reduction in the rate of diabetic foot ulcers in patients with high-risk diabetic feet using 3D printed insoles compared to standard care. The secondary outcome measures will be improvement in standardised QOL measures. 450 diabetes patients with high-risk feet would be recruited who would be prepared to wear the custom made 3D printed insoles on a regular basis (Intervention group). The control group will be formed of 450 diabetes patients with high-risk feet who will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes (type 1 or 2)
* Aged ≥18
* Peripheral sensory neuropathy assessed by 10-gram monofilament With
* Signs of abnormal loading as indicated by callus formation or hyperaemia Or
* limb ischaemia as evidenced by intermittent claudication /non-palpable pulses / history of vascular intervention Or
* on renal replacement therapy

Exclusion Criteria:

* Patients currently prescribed with or in need of therapeutic footwear
* Active or history of foot ulcer
* Active Charcot's neuroarthropathy
* History of major operation in the foot including amputation,
* Local / systemic symptoms of infection, severe illness that would make 12 month survival unlikely
* Unable to provide informed consent
* Inability to follow the study instructions (as judged by the recruiting clinician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
The incidence of new ulcer in patients with high-risk diabetic feet is our primary outcome measure | Within 1 year of randomisation
  Ulcer is defined as any new break in the skin of the feet

SECONDARY OUTCOMES:
To compare patient satisfaction at baseline 26, and 52 weeks post randomisation | Within 1 year of randomisation
  standardised questionnaires
To evaluate quality of life using NeuroQoL at baseline, 26, and 52 weeks post randomisation | Within 1 year of randomisation
  standardised questionnaires
Incidence of adverse events relating in the 3D insole group over 52 weeks post randomisation | Within 1 year of randomisation
  AE event recording
New callus formation | Within 1 year of randomisation
  Clinical examination by podiatrists
To evaluate quality of life using EQ-5D-3L at baseline, 26, and 52 weeks post randomisation | Within 1 year of randomisation
  standardised questionnaires
Need for debridement of callus | Within 1 year of randomisation
  Clinical examination by podiatrists

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Nair, FRCP, PhD, Principal Investigator — Countess of Chester Hospital NHS Trust, Chester, UK
Locations (1):
- Countess of Chester NHS Trust, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided